CLINICAL TRIAL: NCT02934451
Title: Dental Malocclusion and Craniofacial Development in OI
Status: Active, not recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: Shriners Hospitals for Children (Other); Hospital for Special Surgery, New York (Other); University of Nebraska (Other); Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other); Children's National Research Institute (Other); University of California, Los Angeles (Other); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Brendan Lee, Professor and Chairman, Baylor College of Medicine
Other Study IDs: H38629
Record Dates: First submitted 2016-10-12; First posted 2016-10-17 (Estimated); Last update posted 2026-01-27 (Actual); Status verified 2025-01

CONDITIONS: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Osteogenesis imperfecta (OI) is a rare inherited disorder that causes bones to break easily. Individuals with osteogenesis imperfecta break bones often and may have other problems, including hearing loss and pain and difficulty getting around. People with moderate to severe OI may also be diagnosed with dentinogenesis imperfecta (DI). DI is characterized by grey or brown teeth that may chip and wear down and break easily. People with DI may also have skull and neck defects. These patients may have severe teeth misalignment resulting in clinically significant chewing problems. Teeth misalignment in OI is very hard to treat because of the quality and quantity of bone. The overall goal of this study is to improve dental health to improve the quality of life of people with OI.

DETAILED DESCRIPTION:
Investigators will look at dental health in people with OI and will describe teeth misalignment and head and neck defects in individuals with moderate to severe Osteogenesis Imperfecta (OI).

Investigators will look at results from the Longitudinal study of OI to complete the study evaluations. Several x-rays will be performed for this study. Participants will have a 3D scan of the mouth and a Cone Beam CT scan of the jaw at a baseline visit and at 3 years after the baseline visit. These study visits can be at the same time as the Longitudinal Study of OI study visits.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with Clinical diagnosis of OI other than OI type I
* Individuals 10 years or older
* Participant of the Brittle Bone Disease (BBD) Longitudinal Study (7701)

Exclusion Criteria:

* Individuals who cannot be correctly positioned for valid radiographic analysis (e.g., due to severe scoliosis or short neck secondary to basilar invagination)
* Women who are pregnant

Ages: 10 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with Severe OI
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Teeth Misalignment | 5 years
  Measure teeth misalignment in individuals with moderate to severe OI using scans of the teeth.

SECONDARY OUTCOMES:
Neck Defects | 5 years
  Determine neck defects in individuals with moderate to severe OI using scans of the neck and jaw.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Retrouvey, D.M.D., Study Chair — McGill University; Reid Sutton, M.D., Study Chair — Baylor College of Medicine; Frank Rauch, M.D., Study Chair — Shriners Hospital for Children
Locations (3):
- United States (2):
  - University of California Los Angeles, Los Angeles, California
  - Baylor College of Medicine, Houston, Texas
- Shriners Hospital for Children, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
The clinical information collected for this study will be stored in a computer database at the Data Management and Coordinating Center at the University of South Florida in Tampa, FL and also sent to a Federal data repository. A data repository provides a way for researchers to store the information collected during the research study for future research studies. The data management center uses several layers of protection for the clinical data stored in its computer database. It meets all of the local and federal security requirements for research datacenters. Information is stored only using a study identification number. Only the investigators and the study staff who collect and enter study data will have access to the key which links the identification number to the participant.